CLINICAL TRIAL: NCT01296672
Title: Improving Prostate Biopsy Efficiency: The Finasteride Challenge Test
Brief Title: 3 Month Finasteride Challenge Test Can Significantly Improve the Performance of Screening for Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: ROI 10-352H; R01CA138627 (NIH)
Record Dates: First submitted 2011-02-03; First posted 2011-02-15 (Estimated); Results first posted 2017-09-08 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
Keywords: Finasteride; Placebo; Prostate cancer; Prostate Specific Antigen (PSA); Men at intermediate risk of prostate cancer; Men scheduled for prostate biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Finasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Finasteride (Experimental): Finasteride 5mg tablets every day by mouth for 3 months
  Interventions: Drug: Finasteride
- Placebo (Placebo Comparator): Placebo 5mg tablet every day by mouth for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Finasteride — Finasteride 5mg every day by mouth for 3 months
  Other Names: Proscar®; Propecia®
  Arms: Finasteride
Drug: Placebo — Placebo every day by mouth for 3 months
  Arms: Placebo

SUMMARY:
The investigators will propose a novel method to improve prostate cancer screening with PSA, using a 3-month treatment with finasteride, a drug used to treat Benign Prostatic Hyperplasia (BPH) and proven to reduce a man's risk of developing prostate cancer. The investigators will also examine three additional promising tests that may further improve diagnosis of prostate cancer.

DETAILED DESCRIPTION:
The primary goal of this proposal is to determine if a 5-alpha reductase 'challenge' improves screening performance of PSA and DRE in men who are scheduled for prostate biopsy. Currently a higher PSA level leads to a recommendation for prostate biopsy, causing hundreds of thousands of unnecessary biopsies annually in the U.S. We will show that a three-month treatment with finasteride for men with high PSA levels will better predict the man who should have a prostate biopsy. PSA performance after finasteride 'challenge' will also be compared with new tests for prostate cancer. Finasteride is supplied by Merck and Company, Incorporated.

ELIGIBILITY:
Inclusion Criteria:

1. Risk of prostate cancer 20-60% calculated with the on-line Prostate Cancer Prevention Trial (PCPT) prostate cancer risk calculator. (www.prostate-cancer-risk-calculator.com). PSA value must be obtained within 3 months prior to study entry. A description of the frequency of these individuals in the population is provided in Specific Aim 2
2. Patient has been recommended to undergo and plans to have a prostate biopsy.
3. Patient is willing to delay prostate biopsy for a 3-month finasteride vs placebo treatment.
4. No allergy to finasteride or other five alpha reductase inhibitors.
5. Patient is willing to take finasteride vs placebo 5 mg orally daily for 3-month treatment period.
6. Age 55 or older. (This age is selected as the PCPT risk calculator is only valid for this age range.)

Exclusion Criteria:

1. Risk of cancer greater than 60% or less than 20%.
2. Prior history of prostate cancer.
3. Prior treatment with finasteride or dutasteride in the past 6 months
4. Younger than age 55.

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2011-02; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Hernandez, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, Medical Arts and Research Center, San Antonio, Texas, United States

REFERENCES:
- [Derived] Hernandez J, Gelfond J, Goros M, Liss MA, Liang Y, Ankerst D, Thompson IM Jr, Leach RJ. The effect of 3-month finasteride challenge on biomarkers for predicting cancer outcome on biopsy: Results of a randomized trial. PLoS One. 2018 Oct 9;13(10):e0204823. doi: 10.1371/journal.pone.0204823. eCollection 2018. PMID 30300367

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Finasteride | Placebo
Started | 306 | 77
Completed | 233 | 59
Not Completed | 73 | 18
Not completed — Lost to Follow-up | 73 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Finasteride | Placebo | Total
Number analyzed (Participants) | 306 | 77 | 383
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [61 to 68] | 66 [61 to 68] | 65 [61 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 306 | 77 | 383
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Non-Hispanic white | 125 | 31 | 156
  Race: Non-Hispanic black | 42 | 12 | 54
  Race: Hispanic | 134 | 34 | 168
  Race: Other race | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 306 | 77 | 383
Prostate Specific Antigen [Median (Inter-Quartile Range); unit: ng/ml] | 5.2 [4.3 to 6.6] | 5.3 [4.5 to 6.7] | 5.2 [4.3 to 6.6]

OUTCOME MEASURES:

1. Primary Outcome: Pre/Post Ratio PSA Area Under the Curve (AUC)
Description: Pre/Post Ratio prediction area under the receiver operating characteristics curve (AUC) for subjects taking finasteride 5mg every day for 3 months. Measurements of PSA are measured from Baseline until 3 months.
Time Frame: Reported at 90-days: assessment at baseline, 1 month, 2 months and 3 months
Population: Patients with biopsy
Measure: Number (95% Confidence Interval); unit: Ratio
Groups:
- Finasteride; Placebo: PSA Ratio AUC
Arm/Group | Finasteride | Placebo
Number analyzed (Participants) | 233 | 59
Ratio | 0.57 [0.45 to 0.6] | 0.61 [0.46 to 0.76]

2. Secondary Outcome: PCA3 (Prostate Cancer Antigen 3)Score AUC
Description: Area under the Receiver Operating Characteristic Curve (ROC-AUC) of the PCA3 (Prostate Cancer Antigen 3) to detect difference in PSA decline between cases and controls (non-cases)
Time Frame: Reported at 90 days: assessed at baseline, 30 days, 60 days and 90-day
Population: Receiving biopsy
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Finasteride | Placebo
Number analyzed (Participants) | 233 | 59
ratio | 0.65 [0.58 to 0.72] | 0.84 [0.73 to 0.96]

3. Secondary Outcome: T2:ERG ( A Gene on Chromosome 21q22.2 That Encodes an Androgen-regulated Transmembrane Serine Protease Ratio to Estrogen Related Gene) Score AUC
Description: Area Under the Receiver Operating Characteristic Curve (ROC-AUC) of the T2:ERG ( A Gene on Chromosome 21q22.2 That Encodes an Androgen-regulated Transmembrane Serine Protease Ratio to Estrogen Related Gene) Score to Predict the Risk of Prostate Cancer
Time Frame: Reported at 90 days: assessed at baseline, 30 days, 60 days, and 90 days
Population: Receiving biopsy
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | Finasteride | Placebo
Number analyzed (Participants) | 233 | 59
Ratio | 0.62 [0.55 to 0.69] | 0.62 [0.47 to 0.76]

ADVERSE EVENTS:
Arm/Group | Finasteride | Placebo
All-Cause Mortality (participants affected / at risk) | 0/306 | 0/77
Serious Adverse Events (participants affected / at risk) | 3/306 | 1/77
Other Adverse Events (participants affected / at risk) | 7/306 | 6/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finasteride (N=306) | Placebo (N=77)
fulgurated skin lesions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Skin Lesions/tags with itching--fulgurated
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) — "prob" palipitations" heart fluttering X2 seconds
Dizziness (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Morning dizziness while in bed and better when gets out of bed
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Severe abdominal pain
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Finasteride (N=306) | Placebo (N=77)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Decreased libido (Reproductive system and breast disorders) | 3 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Itch (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Stent placement (Vascular disorders) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less